CLINICAL TRIAL: NCT02371239
Title: SIT LESS 2: Effect of Sitting Less on Glucose Regulation in People With Diabetes Mellitus Type 2
Acronym: SIT LESS 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 13-2-050; NL45498.068.13 (Registry Identifier: Medical Ethical Committee Maastricht University Hospital / University of Maastricht)
Record Dates: First submitted 2015-01-22; First posted 2015-02-25 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes
Keywords: Glucose regulation; Glucose; Lipids
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sitting regime (Experimental): The subjects will follow the sitting regime during four days. Each day: 14 hours sitting, 1 hour walking and 1 hour standing for daily care and 8 hours sleeping or lying.
  Interventions: Behavioral: Physical activity intervention
- Sit Less regime (Experimental): Subjects will follow the sit less regime during four days. Each day will consist of 3 hours walking, 4 hours standing, 9 hours sitting and 8 hours sleeping or lying. The additional 2 hours of walking and 3 hours of standing, compared to the sitting regime, will be done in a minimum of four bouts with a time interval of > 1 hour. The subjects will be instructed to walk on a slow pace. i.e. 2-3 km/h, which is comparable to walking during shopping, walking to the office etc.
  Interventions: Behavioral: Physical activity intervention
- Exercise regime (Experimental): Subjects will follow the exercise regime during four days. Each day will consist of 13 hours and 15 minutes sitting, ± 45 minutes supervised cycling on an ergometer, 1 hour walking and 1 hour standing for daily care and 8 hours sleeping or lying.
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention

SUMMARY:
Introduction: Changes in lifestyle are responsible for an important part of the type 2 diabetes epidemic of the last decennia. Current guidelines for physical activity focus mainly on high energy expenditure advising 30 minutes per day moderate to vigorous physical activity (most often physical exercise). Recent studies suggest that sitting has negative metabolic effects independent of the time spent exercising (Duvivier et al. PLOS ONE 2013).

Low intensity physical activity (LIPA) -such as walking and standing- has been suggested to be an alternative to decrease the hyperglycaemic effect of sitting. Compared to exercise, LIPA might be a more feasible strategy. But, it remains to be determined whether reducing sitting time by replacing it by LIPA, results in lower 24 hour blood glucose levels and less blood glucose fluctuations (glycaemic variability) in type 2 diabetes patients and whether these effects are independent of the increase in energy expenditure

Methods: The study population will involve 19 people with type 2 diabetes (BMI: 25-35 kg/m2) who perform no, or only little, exercise and who are treated with diet only or with oral blood glucose lowering medication. They will perform three regimes of each four days: 1) a sitting regime, 2) an exercise regime and a 3) sit less regime. Daily energy expenditure of the exercise regime will be identical to that of the sit less regime. Sitting, walking and standing will be objectively measured by a 24 hour physical activity monitor. The energy spent during exercise will be standardised and quantified by using a bicycle ergometer; energy intake will be standardised as well. During each regime blood glucose will be measured with a 24 hour continuous glucose sensor.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men and women: 40-75 years old
* Diabetes mellitus type 2, developed after the age of 40 years old
* Treatment with diet or oral blood glucose lowering medication (metformin and/or SU-derivatives and/or DPP-IV inhibitors)
* HbA1c: < 10%
* BMI: 25.0 - 35.0 kg/m2
* Maximum 2.5 hours of MVPA per week (during last 3 months)
* Internet availability on a daily basis

Exclusion Criteria:

* Pregnancy or intention of becoming pregnant
* Alcohol use: > 2 units per day (during the last 3 months)
* Experimental drug use (during the last 3 months)
* Use of insulin, corticosteroids, vitamin K antagonists and immunosuppressive drugs in the last 3 months
* Triglyceride level > 10.0 mmol/L
* Fasting plasma glucose level > 10 mmol/L
* Heart failure NYHA 3 or higher
* Angina pectoris or signs of cardiac ischemia during exercise testing
* COPD Gold 3 or higher
* Glomerular filtration rate (GFR) < 30 ml/min
* Diagnosis of active cancer (not cancer in the past that is cured)
* Diabetes mellitus type 1
* Intermittent claudication with a walking distance < 500 meter
* Not able to cycle for ± 45 minutes, as judged from the incremental exhaustive exercise bicycle-ergometer test at Visit 1
* Based on historical information not able to walk for 3 hours per day and stand for 4 hours per day
* Mental or physical disability which makes physical activity not possible
* Participation in a clinical trial with medication use (in the last 3 months)
* Severe loss of vision
* Active foot ulcer or venous leg ulcer

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Mean 24 hour glucose concentration | during the last 24 hours of an activity regime

SECONDARY OUTCOMES:
Total duration (minutes) of hyperglycaemia (glucose > 10 mmol/L) | during the last 24 hours of an activity regime
Mean 24 hour glucose concentration | during a whole activity regime
Total duration of hyperglycaemia (glucose > 10 mmol/L) | during a whole activity regime
Area under the curve of hyperglycaemia (glucose > 10 mmol/L) | during the last 24 hours of an activity regime
Glucose variability measured as SD divided by mean | the last 24 hours of each regime
Total duration of hypoglycaemia (glucose ≤ 3.9 mmol/L) | during a whole activity regime
Fasting total cholesterol | one day after each activity regime
Non-HDL cholesterol | one day after each activity regime
HDL cholesterol | one day after each activity regime
LDL cholesterol | one day after each activity regime
Triglycerides | one day after each activity regime
Apolipoprotein B | one day after each activity regime
Apolipoprotein A | one day after each activity regime
Free fatty acids | one day after each activity regime
Fasting glucose | one day after each activity regime
Fasting insulin | one day after each activity regime
Fasting C-peptide | one day after each activity regime
Fasting CRP | one day after each activity regime
Fasting IL-6 | one day after each activity regime
Fasting IL-1 | one day after each activity regime
Homeostatic model assessment 2 (HOMA2) | one day after each activity regime
  to assess insulin sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaas C Schaper, MD PhD, Principal Investigator — Maastricht University Hospital
Locations (1):
- Human Movement Science, Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Duvivier BM, Schaper NC, Bremers MA, van Crombrugge G, Menheere PP, Kars M, Savelberg HH. Minimal intensity physical activity (standing and walking) of longer duration improves insulin action and plasma lipids more than shorter periods of moderate to vigorous exercise (cycling) in sedentary subjects when energy expenditure is comparable. PLoS One. 2013;8(2):e55542. doi: 10.1371/journal.pone.0055542. Epub 2013 Feb 13. PMID 23418444
- [Derived] Duvivier BM, Schaper NC, Hesselink MK, van Kan L, Stienen N, Winkens B, Koster A, Savelberg HH. Breaking sitting with light activities vs structured exercise: a randomised crossover study demonstrating benefits for glycaemic control and insulin sensitivity in type 2 diabetes. Diabetologia. 2017 Mar;60(3):490-498. doi: 10.1007/s00125-016-4161-7. Epub 2016 Nov 30. PMID 27904925
- See also: Related Info — http://www.plosone.org/article/metrics/info%3Adoi%2F10.1371%2Fjournal.pone.0055542